CLINICAL TRIAL: NCT05154123
Title: A Phase 1, Open-Label Study to Evaluate the Effect of AT-527 on the Pharmacokinetics of Rosuvastatin in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Rosuvastatin and AT-527 (R07496998)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT-03A-012
Record Dates: First submitted 2021-11-16; First posted 2021-12-10 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2021-10

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — AT-511; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AT-527 + rosuvastatin (simultaneous) n=14 (Experimental)
  Interventions: Drug: Drug: AT-527 + rosuvastatin
- AT-527 + rosuvastatin (staggered) n=14 (Experimental)
  Interventions: Drug: AT-527 + rosuvastatin

INTERVENTIONS:
Drug: Drug: AT-527 + rosuvastatin — * Day 1: A single dose of rosuvastatin will be administered.
  * Day 8: A single dose of AT-527 and rosuvastatin will be co-administered.
  Other Names: AT-527 is also know as R07496998
  Arms: AT-527 + rosuvastatin (simultaneous) n=14
Drug: AT-527 + rosuvastatin — * Day 1: A single dose of rosuvastatin will be administered.
  * Day 8: A single staggered dose of AT-527 and rosuvastatin will be administered (2 hours later)
  Other Names: AT-527 is also know as R07496998
  Arms: AT-527 + rosuvastatin (staggered) n=14

SUMMARY:
Drug-drug interaction study of rosuvastatin and AT-527 (R07496998)

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug
* Females must have a negative pregnancy test at Screening and prior to dosing
* Minimum body weight of 50 kg and body mass index (BMI) of 18-29 kg/m2
* Willing to comply with the study requirements and to provide written informed consent

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2
* Abuse of alcohol or drugs
* Use of other investigational drugs within 28 days of dosing
* Concomitant use of prescription medications, or systemic over-the-counter medications
* Other clinically significant medical conditions or laboratory abnormalities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of co-administration of AT-527 on the single-dose pharmacokinetics (PK) of rosuvastatin | Day 1, Day 8
  Maximum plasma concentration (Cmax)
To evaluate the effect of co-administration of AT-527 on the single-dose pharmacokinetics (PK) of rosuvastatin | Day 1, Day 8
  Area under the concentration-time curve (AUC)
To determine the effect of a staggered dose of AT-527 administered 2 hours before rosuvastatin on the PK of rosuvastatin | Day 1, Day 8
  Area under the concentration-time curve (AUC)
To determine the effect of a staggered dose of AT-527 administered 2 hours before rosuvastatin on the PK of rosuvastatin | Day 1, Day 8
  Maximum plasma concentration (Cmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Québec, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No